CLINICAL TRIAL: NCT01848808
Title: The Effect of Wobenzym PS on Inflammation
Acronym: WO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Atrium Innovations (Industry)
Responsible Party: Principal Investigator, Benoit Lamarche, PhD, Laval University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: INAF-2012-076
Record Dates: First submitted 2013-05-03; First posted 2013-05-08 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Sub-clinical Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wobenzym PS (Experimental): During the 4-week of the Wobenzym supplementation, participants will take 6 tablets of Wobenzym: 2 tablets 3 times daily at least 45 minutes before meal.
  Interventions: Dietary Supplement: Wobenzym PS
- Placebo (Placebo Comparator): During the 4-week of placebo phase, participants will take 6 tablets of placebo: 2 tablets 3 times daily at least 45 minutes before meal.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Wobenzym PS
  Arms: Wobenzym PS
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The general objective of this project is to examine the impact of Wobenzym PS supplementation on blood markers of inflammation and inflammation gene expression in volunteers with sub-clinical inflammation.

The study will be undertaken according to a double-blind, cross over, randomized, placebo controlled design. The study will involve men and women with subclinical inflammation (n=24). Eligible subjects will have blood CRP >1 mg/L and <10 mg/L and will be in good health. The impact of Wobenzym PS on inflammation (vs. placebo) will be assessed by comparing the blood fasting concentrations and whole blood gene expression of anti- and pro-inflammatory proteins before and after the 4-week supplementation (Wobenzym and placebo). The two 4-week supplementation will be separated by a 4-week wash out period.

DETAILED DESCRIPTION:
Inflammation is being increasingly recognized as key etiological factor in the development of atherosclerosis and subsequent cardiovascular disease (CVD). This pro-atherogenic state is strongly correlated and often found co-segregating among individuals with obesity and metabolic syndrome. There is increasing evidence to support the use in clinical practice of these novel markers of atherosclerosis and CVD risk. C-reactive protein (CRP) has been used extensively as a non-specific marker of acute phase response in clinical practice for decades. More recently, CRP has also been proposed to be a new cardiovascular biomarker of atherosclerosis and its complications. Studies that have investigated the predictive value of sub-acute CRP levels have been relatively consistent in showing that individuals with high hsCRP (high-sensitivity C-reactive protein) levels (>3.0 mg/L) were at greater risk of CVD compared to individuals with lower (<1.0 mg/L) hsCRP levels, independent of gender and plasma cholesterol concentrations. Wobenzym is an enzyme formula primarily recommended for the treatment of pain and inflammation associated with musculoskeletal disorders. Several studies in the areas of arthritis and post-surgery have reported the acute anti-inflammatory effects of Wobenzym in terms of changes in CRP. Whether Wobenzym plays a role in managing sub-acute inflammation as well remains to be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18-75 years
* Subclinical inflammation (CRP levels > 1 mg/L and < 10 mg/L)

Exclusion Criteria:

* Hypersensitivity to Wobenzym PS constituents
* Severe congenital or acquired coagulation disorders (e.g. haemophilia, in dialysis patients)
* Severe liver damage
* Prior to surgical operations
* Any clinical signs or laboratory evidence for severe inflammatory, endocrine, renal/pulmonary, neurological, cardiovascular, metabolic, haematological, or psychiatric condition, which in the Investigator's opinion contraindicates a 4-week course of Wobenzym PS use
* Active malignancy of any type or history of a malignancy within the last five years other than basal cell carcinoma.
* Any active gastrointestinal disease
* Use of anticoagulants or thrombocyte aggregation inhibitors, chemotherapeutic agents, antibiotics, medication for lipids, diabetes, hypertension, inflammation, autoimmune diseases, mood disorders
* Use of NSAID (nonsteroidal antiinflammatory drug) within 1 month of entering the study
* Excessive alcohol consumption (more than two drinks by day for men, one for women) and active alcoholism; smoking; drug use and history of drug abuse; supplements or natural products consumption during the study
* Pregnant or breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in the expression of anti- and pro-inflammatory genes in total blood RNA from white blood cells (WBC) | At the end of the two 4-weeks supplementation (week 4 and week 12)

SECONDARY OUTCOMES:
Change in blood levels of anti- and pro-inflammatory markers | At the end of the two 4-weeks supplementation (week 4 and week 12)

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Lamarche, PhD, Principal Investigator — Laval University
Locations (1):
- Institute of nutrition and functionnal foods, Québec, Quebec, Canada